CLINICAL TRIAL: NCT07378995
Title: The Effect of Therapeutic Play Applied Before Intramuscular Injection on Fear, Anxiety and Pain in Pre-school Children
Brief Title: The Effect of Therapeutic Play Applied Before Intramuscular Injection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ARZU SARIALİOĞLU, Associate professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 30.2.ATA.0.01.0
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Child, Only; Fear; Pain
MeSH Terms: conditions — Pain | interventions — Play Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- therapeutic play (Experimental): Children in the intervention group will be introduced to therapeutic toy dolls and will be educated on what to do with them. Prior to the training, children will be informed about the importance of intramuscular injections and how they are administered. The reasons for the injection and how it is administered will be explained in detail.
  Participants will be shown the steps involved in intramuscular injection. Using a toy doll, the steps of intramuscular injection will be demonstrated step by step, and the children will practise applying these steps. During the training, children will be told in detail how to administer injections carefully, where the injection should be given, and how to perform the injection correctly. At the end of the training, children will successfully perform the intramuscular injection procedure. The injection will then be administered to the children by the same nurse who received training from the research team.
  Interventions: Behavioral: therapeutic play
- control (No Intervention): Children in the control group will receive the IM injection at the clinic using routine practice methods.The injection will be administered by the same nurse trained by the research team.

INTERVENTIONS:
Behavioral: therapeutic play — Children in the intervention group will be introduced to therapeutic toy dolls and will be educated on what to do with them. Prior to the training, children will be informed about the importance of intramuscular injections and how they are administered. The reasons for the injection and how it is administered will be explained in detail.
  Participants will be shown the steps involved in intramuscular injection. Using a toy doll, the steps of intramuscular injection will be demonstrated step by step, and the children will practise applying these steps. During the training, children will be told in detail how to administer injections carefully, where the injection should be given, and how to perform the injection correctly. At the end of the training, children will successfully perform the intramuscular injection procedure. The injection will then be administered to the children by the same nurse who received training from the research team.
  Arms: therapeutic play

SUMMARY:
This research aims to evaluate the effectiveness of a therapeutic toy doll developed to reduce the levels of fear, anxiety and pain experienced by children aged 4-6 during intramuscular injection procedures.

Children, especially at an early age, show great sensitivity towards medical procedures, and these processes can often cause pain, anxiety and fear. This research aims to evaluate the effectiveness of a therapeutic toy doll developed to reduce the levels of fear, anxiety and pain experienced by children aged 4-6 during intramuscular injection procedures. Children, especially at an early age, show great sensitivity to medical procedures, and these processes can often cause pain, anxiety, and fear. This research aims to discover methods of managing and improving children's responses to medical procedures through therapeutic games.

This study, to be conducted at the Emergency Department of Atatürk University Research Hospital in Erzurum, will be carried out using a randomised controlled design. Participants will be randomly assigned to intervention and control groups. Children in the intervention group will prepare using the therapeutic toy doll, while children in the control group will receive an intramuscular injection at the clinic using routine application methods.

Data collection tools will include the Socio-demographic Information Form, the Children's Fear Scale (CFS), the Children's Anxiety Scale-State (CAS-D), and the Wong-Baker Facial Expression Rating Scale.

DETAILED DESCRIPTION:
This study, to be conducted at the Emergency Department of Atatürk University Research Hospital in Erzurum, will be carried out using a randomised controlled design. Participants will be randomly assigned to intervention and control groups. Children in the intervention group will prepare using the therapeutic toy doll, while children in the control group will receive an intramuscular injection at the clinic using routine application methods.

Data collection tools will include the Socio-demographic Information Form, the Children's Fear Scale (CFS), the Children's Anxiety Scale-State (CAS-D), and the Wong-Baker Facial Expression Rating Scale.The original value of the research lies in the development of a therapeutic toy doll for intramuscular injection and in evaluating the effect of this therapeutic toy doll on children undergoing the injection procedure through therapeutic play. The therapeutic toy doll aims to familiarise children with the injection process and make them find this process less frightening, thereby experiencing less stress during the actual injection.

This approach aims to reduce children's fear, anxiety, and pain levels towards medical procedures and help them develop a positive outlook.

The expected results of the research indicate that children who receive injections with the therapeutic toy doll may experience a significant reduction in their levels of fear, anxiety, and pain. The therapeutic toy doll may help children cope with challenging medical situations and enable them to interpret their experiences with healthcare services in a more positive manner. The research findings will contribute to the development of new strategies for medical procedures in paediatric care that result in less fear, pain, and anxiety. Healthcare professionals and families will gain practical and effective tools to facilitate children's adaptation to medical procedures.

This research will contribute to raising standards in children's healthcare services and offer innovative approaches that enable children to have more positive health experiences.

This research aims to present innovative approaches that will enable the raising of standards in children's health services and allow children to have more positive health experiences.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-6 years,
* Those who will receive intramuscular injections,
* Those who have been prescribed Desefin flk 1x1 IM,
* Children whose parents have given consent will be included in the study.

Exclusion Criteria:

* Those experiencing pain,
* Those with hearing problems and communication barriers,
* Those with chronic illnesses,
* Those with mental and physical disabilities,
* Those who have taken analgesics within the last 6 hours,
* Children who have previously been hospitalised will not be included in the study.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Child Fear Scale | 1 year
  The scale was developed by McMurty et al. to measure fear in children undergoing painful medical procedures. Its validity and reliability in Turkish were established by Gerçeker et al. The scale features five distinct facial expressions, ranging from no fear/anxiety at one end to very intense fear/anxiety at the other, and is scored on a scale of 0 to 4. 0 indicates no fear/anxiety, while 4 indicates extreme fear and anxiety
Child Anxiety Scale-State | 1 year
  The scale developed by Ersig et al. has been validated and tested for reliability in Turkish by Özalp Gerçeker et al. The CAS-D resembles a thermometer with a bulb at the bottom and horizontal lines extending upwards at intervals. In this scale, which is aimed at children aged four to ten, children are instructed to "think of all your anxious or nervous feelings as being in the bulb or lower part of the thermometer. If you feel a little anxious or nervous, your feelings may rise a little higher on the thermometer. If you are very, very anxious or nervous, your feelings may go all the way to the top. Place a line on the thermometer to show how anxious or nervous you are." To measure state anxiety (CAS-D), the child is asked to mark how they feel 'right now'. A transparent ruler marked in ½-point increments is placed over the child's rating, and the ½-point increment is then rounded to the nearest number. The score can range from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Nursing of Faculty, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.